CLINICAL TRIAL: NCT00185289
Title: Multi-center , Open, Uncontrolled Study to Investigate the Efficacy and Safety of a 4 Phasic Oral Contraceptive SH T00658 in a 28-day Regimen for 20 Cycles in Healthy Female Volunteers
Brief Title: Study to Investigate Efficacy and Safety of a New Oral Contraceptive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare AG
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 91191; EudraCT: 2004-002098-22; 306660
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Contraception

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658K)

INTERVENTIONS:
Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658K) — per cycle (28 days): Days 1-2: 3.0 mg EV; Days 3-7: 2.0 mg EV + 2.0 mg DNG; Days 8-24: 2.0 mg EV + 3.0 mg DNG; Days 25-26: 1.0 mg EV; Days 27-28: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of a new 4-phasic preparation in the prevention of pregnancies in a large group of volunteers.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Any condition that might interfere the outcomes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1392 (Actual)
Dates: Start 2004-04; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Number of unintended pregnancies | 20 treatment cycles each consisting of 28 days and follow-up period of 14 days

SECONDARY OUTCOMES:
Adverse event collection | 20 treatment cycles each consisting of 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (50):
- Austria (18):
  - Dr. Max Stiglbauer, Wiener Neustadt, Lower Austria
  - Praxis Dr. Langer, Fürstenfeld, Styria
  - Dr. Meusburger, Wolfurt, Vorarlberg
  - Landeskrankenhaus Bregenz, Bregenz
  - Dr. Roswitha Wessely, Graz
  - Institut für Hormonstörungen und Kinderwunsch, Graz
  - Praxis Dr. Gudrun Lorenz-Eberhard, Graz
  - Praxis Dr. Hannes Kahr, Graz
  - Universitätsklinikum Innsbruck, Innsbruck
  - Dr. Peter Mayr, Kufstein
  - Dr. Michaela Boeckl, Salzburg
  - Dr. Sigrid Schmidl-Amann, Sankt Pölten
  - Dr. Guenther Heytmanek, Vienna
  - Dr. Ewald Boschitsch, Vienna
  - Dr. Brigitte Wiesenthal, Vienna
  - Allgemeines Krankenhaus der Stadt Wien Universitätskliniken, Vienna
  - Dr. Wolfgang Bartl, Vienna
  - Dr. Walter Paulik, Zeltweg
- Germany (27):
  - Praxis Hr. Dr. A. Soder, Ettlingen, Baden-Wurttemberg
  - Praxis Hr. Dr. U. Kohoutek, Karlsruhe, Baden-Wurttemberg
  - Praxis Hr. Dr. L. Weihe, Ansbach, Bavaria
  - Praxis Hr. Dr. D. Rautenberg, Hamburg, Hamburg
  - Frauenarztpraxis Dr. med. Wolfram Brach, Dietzenbach, Hesse
  - Praxis Hr. Dr. Werner Göttker-Schnetmann, Frankfurt am Main, Hesse
  - Praxis Dr. S. El Tobgui-Jensen, Frankfurt am Main, Hesse
  - Praxis Dr. S. Clauss-Hoffmann, Frankfurt am Main, Hesse
  - Praxis Hr. Dr. P. Schwaner, Frankfurt am Main, Hesse
  - Praxis Dr. Kindt, Langen, Hesse
  - Praxis Fr. Dr. J. Tyagi, Mühlheim am Main, Hesse
  - Praxis Hr. Dr. H. Zabel, Bovenden, Lower Saxony
  - Praxis Hr. Dr. K. Brauns, Hamelin, Lower Saxony
  - Praxis Hr. Dr. K. Greven, Hanover, Lower Saxony
  - Praxis Hr. Dr. H. Frommeyer, Osnabrück, Lower Saxony
  - Frauenarztpraxis Dr. Schoenberg, Rheine, North Rhine-Westphalia
  - Praxis Fr. I. Gröger, Wurzen, Saxony
  - Praxis Hr. H. Thelen, Jessen, Saxony-Anhalt
  - Frauenarztpraxis Dr. med. Gabriele Weinreich, Magdeburg, Saxony-Anhalt
  - Dinox GmbH Berlin, Berlin, State of Berlin
  - Charité Campus Benjamin Franklin, Berlin, State of Berlin
  - Frauenarztpraxis Fr. Dr. S. Gramatte, Berlin, State of Berlin
  - Praxis Fr. Dr. B. Wernecke, Berlin, State of Berlin
  - Praxis Fr. Dr. I. Hannig, Berlin, State of Berlin
  - Praxis Fr. Dr. K. Maar, Berlin, State of Berlin
  - Praxis Hr. Dr. R. Etzrodt, Gera, Thuringia
  - Frauenarztpraxis Fr. Dr. H. Schlegel, Saalfeld, Thuringia
- Spain (5):
  - USP Institut Universitari Dexeus, Barcelona, Barcelona
  - Diatros Gava- Centre Assistencial Ntra. Sra. de Burgues, Gavà, Barcelona
  - Hospital Universitario MAterno Infantil de Canarias, Las Palmas, Gran Canaria
  - Instituto Palacios de Salud y Medicina de la Mujer, Madrid
  - Complejo Hospitalario Ntra. Sra. de Valme, Seville